CLINICAL TRIAL: NCT05898776
Title: Safety of 10°C Lung Preservation vs. Standard of Care: A Multi-Centre Prospective Non-Inferiority Trial
Brief Title: 10°C vs 4°C Lung Preservation RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Medical University of Vienna (Other); Vanderbilt University (Other); Puerta de Hierro University Hospital (Other); University of California, San Francisco (Other); Centre Hospitalier Universitaire Vaudois (Other); Mayo Clinic (Other); St Vincent's Hospital, Sydney (Other); University of Texas Southwestern Medical Center (Other); Corewell Health West (Other); University of Miami (Other); University Hospital of Leuven Leuven (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other); University Hospital, Zürich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-5909
Record Dates: First submitted 2023-05-31; First posted 2023-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Lung Transplant; Organ Preservation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 10°C lung preservation (Experimental)
  Interventions: Device: Lung transplantation after 10°C donor lung preservation
- Standard lung preservation (Active Comparator)
  Interventions: Device: Lung transplantation after standard ice cooler donor lung preservation

INTERVENTIONS:
Device: Lung transplantation after 10°C donor lung preservation — When suitable donor lungs become available for a, eligible, consented recipient and meet criteria to go straight to transplantation, the lungs randomized to 10°C preservation will be stored, transported and preserved in the X°Port Lung Transport Device (Traferox Technologies Inc.) until implant with a maximum time of 12 hours between the donor and recipient surgeries.
  Arms: 10°C lung preservation
Device: Lung transplantation after standard ice cooler donor lung preservation — When suitable donor lungs become available for a, eligible, consented recipient and meet criteria to go straight to transplantation, the lungs randomized to standard preservation will be will be stored, transported and preserved in an ice cooler (~4°C, standard of care) until implant with a maximum time of 6 hours between the donor and recipient surgeries.
  Arms: Standard lung preservation

SUMMARY:
Despite lung transplantation (LTx) being the most effective treatment for end-stage lung disease, its success rate is lower than that of other solid organ transplantations. Primary graft dysfunction (PGD) is the most common post-operative complication and a major factor in early mortality and morbidity, affecting ~25% of lung transplant patients. Induced by ischemia reperfusion, PGD represents a severe and acute lung injury that occurs within the first 72 hours after transplantation, and has a significant impact on short- and long-term outcomes, and a significant increase in treatment costs. Any intervention that reduces the risk of PGD will lead to major improvements in short- and long-term transplant outcomes and health care systems.

One of the main strategies to reduce the risk and severity of post-transplant PGD is to improve pre-transplant donor lung preservation methods. In current practice, lung preservation is typically performed by cold flushing the organ with a specialized preservation solution, followed by subsequent hypothermic storage on ice (~4°C). This method continues to be used and applied across different organ systems due to its simplicity and low cost. Using this method for the preservation of donor lungs, the current maximum accepted preservation times have been limited to approximately 6-8h. While the goal of hypothermic storage is to sustain cellular viability during ischemic time through reduced cellular metabolism, lower organ temperature has also been shown to progressively favor mitochondrial dysfunction. Therefore, the ideal temperature for donor organ preservation remains to be defined and should maintain a balance between avoidance of mitochondrial dysfunction and prevention of cellular exhaustion. In addition to that, safe and longer preservation times can lead to multiple advantages such as moving overnight transplants to daytime, more flexibility to transplant logistics, more time for proper donor to recipient matching etc.

Building on pre-clinical research suggesting that 10°C may be the optimal lung storage temperature, a prospective, multi-center, non-randomized clinical trial was conducted at University Health Network, Medical University of Vienna and Puerta de Hierro Majadahonda University Hospital. Donor lungs meeting criteria for direct transplantation and with cross clamp times between 6:00pm - 4:00am were intentionally delayed to an earliest allowed start time of 6:00am and a maximum preservation time from donor cold flush to recipient anesthesia start time of 12 hours. Lungs were retrieved and transported in the usual fashion using a cooler with ice and transferred to a 10°C temperature-controlled cooler upon arrival to transplant hospital until implantation. The primary outcome of this study was incidence of Primary Graft Dysfunction (PGD) Grade 3 at 72h, with secondary endpoints including: recipient time on the ventilator, ICU Length of Stay (LOS), hospital LOS, 30-day survival and lung function at 1-year. Outcomes were compared to a contemporaneous conventionally transplanted recipient cohort using propensity score matching at a 1:2 ratio. 70 patients were included in the study arm. Post-transplant outcomes were comparable between the two groups for up to 1 year. Thus, intentional prolongation of donor lung preservation at 10°C was shown to be clinically safe and feasible.

In the current study design, the investigators will conduct a multi-centre, non-inferiority, randomized, controlled trial of 300 participants to compare donor lung preservation from the time of explant to implant at ~10°C in X°Port Lung Transport Device (Traferox Technologies Inc.) vs a standard ice cooler. When eligible donor lungs become available for a consented recipient, the lungs will be randomized to undergo a preservation protocol using either 10°C (X°Port Lung Transport Device, Traferox Technologies Inc.) or standard of care. The primary outcome of the study is incidence of ISHLT Primary Graft Dysfunction Grade 3 at 72 hours. Post-transplant outcomes will be followed for one year.

ELIGIBILITY:
Donor Inclusion Criteria

* Donation after brain death (DBD) or donation after cardiac death (DCD)
* Donor lungs are suitable to go straight to LTx (i.e., do not need ex vivo lung perfusion (EVLP) assessment)

Donor Exclusion Criteria

* Concerns with organ preservation technique
* Need for EVLP assessment

Recipient Inclusion Criteria

* 18-80 years old
* Primary lung transplantation
* Bilateral lung transplantation

Recipient Exclusion Criteria

* Re-transplantation
* Multi-organ transplantation
* Single lung transplantation
* Participation in a contraindicating trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Primary Graft Dysfunction (PGD) Grade 3 as per International Society for Heart and Lung Transplantation (ISHLT) | 72 hours post-transplant
  PGD is graded on a scale of 0 to 3 based on ISHLT guidelines, where PGD Grade 3 indicates severe primary graft dysfunction.

SECONDARY OUTCOMES:
Incidence of Primary Graft Dysfunction Grade 2-3 as per International Society for Heart and Lung Transplantation | 0 (ICU arrival), 24, 48, and 72 hours post-transplant
  PGD is graded on a scale of 0 to 3 based on ISHLT guidelines, where PGD Grade 3 indicates severe primary graft dysfunction.
Time on ventilator | Index hospitalization (up to 1 year)
Total ICU and hospital length of stay | Index hospitalization (up to 1 year)
Overall survival | 30 days, 1 year post-transplant
Occurrence of acute rejection | 1 year post-transplant
Six minute walk test | 1 year post-transplant
Forced expiratory volume - one second (FEV1 in L) | 1 year post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Wakeam, MD MPH, Principal Investigator — University Health Network, Toronto
Locations (14):
- United States (6):
  - University of California San Francisco, San Francisco, California
  - University of Miami, Coral Gables, Florida
  - Corewell Health Research Institute, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
- St Vincent's Hospital Sydney Limited, Sydney, New South Wales, Australia
- Medical University of Vienna, Vienna, Austria
- University Hospitals Leuven, Leuven, Belgium
- Canada (2):
  - University Health Network (Toronto General Hospital), Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
- Hospital Universitario Puerta de Hierro-Majadahonda, Madrid, Spain
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - University Hospital Zurich, Zurich